CLINICAL TRIAL: NCT02761876
Title: Singida Nutrition and Agroecology Project
Acronym: SNAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Nelson Mandela African Institute of Science and Technology (Unknown); Action Aid Tanzania (Other); Ilonga Agricultural Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1511005983
Record Dates: First submitted 2016-03-11; First posted 2016-05-04 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Participatory education) (Experimental): Participatory education
  Interventions: Behavioral: Mentor farmer training (Malawi); Behavioral: Mentor farmer training (Singida, Tanzania); Behavioral: Mentor farmer visits and facilitation
- Control (No Intervention): Delayed participatory education

INTERVENTIONS:
Behavioral: Mentor farmer training (Malawi) — Mentor farmers, 1 man, 1 woman, from each village will participate in a field visit to and training by existing mentor farmers in Malawi. Only the intervention arm of this study will receive mentor farmer training in Malawi, delayed intervention arm will receive mentor farmer training from farmers participating in the initial intervention in Tanzania.
  Arms: Intervention (Participatory education)
Behavioral: Mentor farmer training (Singida, Tanzania) — Mentor farmers will receive training in Singida, Tanzania on agroecology practices, climate change, nutrition, and gender equality. Intervention villages will receive training in 2016. Delayed intervention villages will receive training in 2019.
  Arms: Intervention (Participatory education)
Behavioral: Mentor farmer visits and facilitation — Mentor farmers will conduct monthly visits to participating households and support the households in conducting experimentation with agroecological practices and/or new behavior regarding nutrition and gender equality. Quarterly meetings among farmers within each village will be held to discuss progress and challenges of household experimentations. Intervention households will receive support and facilitation for approximately 2 years. Delayed intervention households will receive support and facilitation for approximately 6 months after end line survey.
  Arms: Intervention (Participatory education)

SUMMARY:
The purpose of this study is to test if a participatory, agroecological peer farmer-led education intervention can be effective at improving legume production, food security, and infant and young child feeding practices in Singida District, Tanzania.

DETAILED DESCRIPTION:
Approximately 40% of under five children in Tanzania are stunted, with higher levels in rural areas. Our inception research in Singida identified five pressing issues faced by smallholder farmers that may contribute to this high rate of stunting. They are (A) hierarchical, or "top down" farmer education, (B) low soil fertility and little knowledge of agroecological solutions, (C) high levels of gender inequality and high workloads for women, (D) food insecurity and low dietary diversity, and (E) sub-optimal infant and young child feeding. Singida Nutrition and Agroecology Project (SNAP) is a randomized effectiveness trial of a participatory, agroecological peer farmer education intervention. Each intervention village will choose 2 mentor farmers, 1 man and 1 woman, who will participate in a field visit to and training by existing mentor farmers in Malawi and a two week long follow-up and refresher trainings in Tanzania integrating agroecology, climate change, nutrition, and gender equality. Mentor farmers will then conduct monthly visits to participating households and support the households in conducting experimentation with agroecological practices and/or new behaviors regarding nutrition and gender equality. Quarterly meetings among mentor farmers and biannual meeting of participating farmers within each village will be held to discuss progress and challenges of peer education and household experimentations.

ELIGIBILITY:
Inclusion Criteria:

* Are among the most vulnerable, as indicated by food insecurity
* Have a child who will be <= 1 year old in February 2016
* Are farmers who have regular access to the same farms/plots (but they do not need to own the land per se)
* Female headed households are acceptable, so long as not more than half the selected households in the village are female headed (to be able to detect change in gender equity)
* Willing to stay in study for 3 years, i.e. do not plan to move
* Interested in experimenting with new farming techniques

Exclusion Criteria:

* Refuses to take part

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2016-02; Primary Completion 2019-02 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Change in dietary diversity score (mean and proportion of score >4) | Twice a year for the first three years of study (2016, 2017, 2018) and once in the final year (2019)
  As defined by World Health Organization (see Citations), this refers to the number of food groups (out of 7) consumed by children the previous day ."

SECONDARY OUTCOMES:
Change in mean child's height-for-age z-score | Twice a year for the first three years of study (2016, 2017, 2018) and once in the final year (2019)
  According to World Health Organization growth chart
Change in proportion of children who are stunted (HAZ<-2) | Twice a year for the first three years of study (2016, 2017, 2018) and once in the final year (2019)
  According to World Health Organization growth chart
Change in mean child's weight-for-height z-score | Twice a year for the first three years of study (2016, 2017, 2018) and once in the final year (2019)
  According to World Health Organization growth chart
Change in proportion of children who are wasted (WHZ<-2) | Twice a year for the first three years of study (2016, 2017, 2018) and once in the final year (2019)
  According to World Health Organization growth chart
Change in mean Food Insecurity Score | Twice a year for the first three years of study (2016, 2017, 2018) and once in the final year (2019)
  Household Food Insecurity Access Scale (HFIAS)
Change in proportion of households with severe or moderate food insecurity | Twice a year for the first three years of study (2016, 2017, 2018) and once in the final year (2019)
  Household Food Insecurity Access Scale (HFIAS)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel N Bezner Kerr, MS PhD, Principal Investigator — Cornell University; Sera L Young, MA PhD, Principal Investigator — Cornell University; Elias Mtinda, Principal Investigator — Action Aid Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Santoso MV, Bezner Kerr RN, Kassim N, Martin H, Mtinda E, Njau P, Mtei K, Hoddinott J, Young SL. A Nutrition-Sensitive Agroecology Intervention in Rural Tanzania Increases Children's Dietary Diversity and Household Food Security But Does Not Change Child Anthropometry: Results from a Cluster-Randomized Trial. J Nutr. 2021 Jul 1;151(7):2010-2021. doi: 10.1093/jn/nxab052. PMID 33973009